CLINICAL TRIAL: NCT06225934
Title: The Effect of Home Exercise Programs Applied in Cooperation With the Family on the Treatment of Congenital Muscular Torticollis.
Brief Title: The Effect of Home Exercise Programs Applied of Congenital Muscular Torticollis.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Gazi University (Other)
Responsible Party: Principal Investigator, Sinem Erturan, principal investigator, Gazi University
Other Study IDs: muscular torticollis
Record Dates: First submitted 2024-01-17; First posted 2024-01-26 (Actual); Last update posted 2024-01-26 (Actual); Status verified 2024-01

CONDITIONS: Congenital Muscular Torticollis; Family Members
Keywords: Cooperation with the family; Congenital Muscular Torticollis
MeSH Terms: conditions — Congenital torticollis | interventions — Exercise

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- congenital muscular torticollis: Babies diagnosed with congenital muscular torticollis (CMT) who agree to participate in the study and meet the inclusion criteria will be included in the study without using any sample selection method, since it is a single-arm study. The parents of each baby will first be informed about the content of the study and will read and sign the consent form stating that they participate in the study voluntarily.
  Interventions: Behavioral: Exercise and home program to increase lateral flexion and rotation angles

INTERVENTIONS:
Behavioral: Exercise and home program to increase lateral flexion and rotation angles — Suggestions will be made to the parent/caregiver of the baby diagnosed with congenital muscular torticollis (CMT) participating in the study to increase the baby's decreasing lateral flexion and rotation angles, and parents/caregivers will be advised to integrate these suggestions into their daily routine as much as possible.These suggestions; It includes holding-carrying-breastfeeding (feeding) principles, active-passive lateral flexion and active stretching of the child and activities that will increase joint range of motion for the SCM muscle, environmental arrangements, games that enable the development of active symmetrical movements and prone activities. The home program to be implemented by parents/caregivers will continue for 6 weeks. During the evaluations, the demographic characteristics of the babies (gender, gestational age, birth weight, parental information, mother's pregnancy type, pregnancy history, Apgar score, ultrasonography values, etc.) will be recorded.

SUMMARY:
Congenital muscular torticollis (CMT) is the third most common musculoskeletal disorder of infancy, affecting 3.9% to 16% of infants. It develops due to unilateral shortening of the SCM, whether or not there is a mass in the sternocleidomastoid muscle (SCM). CMT is characterized by lateral flexion of the affected SCM to the ipsilateral side and rotation to the contralateral side. Its etiology is not fully known. However, it can be associated with SCM disorder that develops due to birth trauma, prenatal/perinatal compartment syndrome and intrauterine restriction. It has been reported that conditions such as multiple pregnancy, intrauterine stenosis, vascular causes, fibrosis of the peripartum bleeding area, use of forceps at birth, difficult birth, and primary myopathy of SCM increase the possibility of CMT. It is necessary to approach babies diagnosed with CMT with an effective treatment program. The most important and effective of these approaches is to provide the necessary education and an intensive home program to their families, with whom they spend most of their days. By educating the family, on the one hand, the baby will receive regular treatment and the family's communication with the baby will be strengthened, while on the other hand, limitations such as transportation, time and cost will be eliminated. In our study; It was aimed to examine the effectiveness of the home program given in cooperation with the family in babies diagnosed with CMT and to create a new protocol.

DETAILED DESCRIPTION:
Congenital muscular torticollis (CMT) is the third most common musculoskeletal disorder of infancy, affecting 3.9% to 16% of infants. It develops due to unilateral shortening of the SCM, whether or not there is a mass in the sternocleidomastoid muscle (SCM). CMT is characterized by lateral flexion of the affected SCM to the ipsilateral side and rotation to the contralateral side. Its etiology is not fully known. However, it can be associated with SCM disorder that develops due to birth trauma, prenatal/perinatal compartment syndrome and intrauterine restriction. It has been reported that conditions such as multiple pregnancy, intrauterine stenosis, vascular causes, fibrosis of the peripartum bleeding area, use of forceps at birth, difficult birth, and primary myopathy of SCM increase the possibility of CMT. These conditions cause degeneration of SCM fibers, edema in SCM, and fibrosis, as well as the general posture seen in SCM. Although CMT seems to be a condition that only concerns the neck muscles; In later periods, it may cause permanent disorders in body biomechanics such as asymmetry in the use of the upper extremities, delay in gross motor functions, postural disorders such as plagiocephaly and scoliosis, and balance disorders. Therefore, babies diagnosed with CMT should be included in a comprehensive and regular physiotherapy and rehabilitation program from the early period. These programs generally include joint range of motion-stretching exercises for the neck, family education including teaching the principles of holding and carrying, approaches such as microcurrent applications and taping, and in more severe cases, botulinum toxin-A (BOTOX-A) or surgical applications. It is necessary to approach babies diagnosed with CMT with an effective treatment program. The most important and effective of these approaches is to provide the necessary education and an intensive home program to their families, with whom they spend most of their days. By educating the family, on the one hand, the baby will receive regular treatment and the family's communication with the baby will be strengthened, while on the other hand, limitations such as transportation, time and cost will be eliminated. In our study; It was aimed to examine the effectiveness of the home program given in cooperation with the family in babies diagnosed with CMT and to create a new protocol.

In our study; It is aimed to examine the effect of the home program given to babies diagnosed with Congenital Muscular Torticollis (CMT) between the ages of 0-12 months, in cooperation with the family, on the treatment of CMT and to contribute to the literature with this approach that can be used by clinicians by creating a treatment protocol for this.

ELIGIBILITY:
Inclusion Criteria:

* Babies aged 0-12 months with a diagnosis of congenital muscular torticollis (CMT)
* Families who agree to participate in the study will be included in the exercise program

Exclusion Criteria:

* Those who have any neurological risk factors were included in the study,
* Those who are affected by their visual/hearing senses,
* Those who have not been diagnosed with Congenital muscular torticollis (CMT) by a doctor,
* Those who have previously received treatment for the diagnosis of CMT,
* Babies with a history of BOTOX-A/surgery applied to the Sternocleidomastoid (SKM) muscle before treatment will not be included.

Ages: 1 Month to 12 Months | Sex: All
Age Groups: Child
Study Population: Fifteen babies diagnosed with congenital muscular torticollis (CMT) who are between 0-12 months old and agree to participate in the study will be included in the study. Congenital muscular torticollis (CMT) is the third most common musculoskeletal disorder of infancy, affecting 3.9% to 16% of infants. It develops due to unilateral shortening of the SCM, regardless of whether there is a mass in the sternocleidomastoid muscle (SCM). CMT is characterized by lateral flexion of the affected SCM to the ipsilateral side and rotation to the contralateral side.
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2024-01-15 (Actual); Primary Completion 2024-03-15 (Estimated); Study Completion 2024-03-15 (Estimated)

PRIMARY OUTCOMES:
Test Of Sensory Functions In Infants (TSFI) | 1-12 months
  It will be used to evaluate the sensory development of babies. The test is frequently used to evaluate the sensory processing functions of babies aged 4-18 months. It is used to determine whether a baby has a sensory processing problem and to what extent. It consists of 24 items.
Peabody Developmental Motor Scales-2 | 1-12 months
  It is planned to use the Peabody Motor Development Scale-2 (PMDS-2) to evaluate motor development. It is designed to identify developmental delays in children between the ages of 0-72 months. It is used to evaluate children's motor development with separate tests and rating scales for both gross motor skills and fine motor skills.
Hammersmith Infant Neurological Examination (HINE) | 1-12 months
  It is planned to be used for neurological status evaluation. It is a neurological examination consisting of 3 separate parts, standardized for babies aged 2-24 months. It contains a total of 37 items examining neurological status, motor development and behavioral status. The test evaluates cranial nerve function, movements, reflexes, posture and tonus, motor development stages, social orientation, emotional state and alertness. Total score varies between 0-78 points. A higher score indicates that the baby's condition is better.
Arthrodial protractor | 1-12 months
  It is planned to use an arthrodial protractor to determine the lateral flexion and rotation range of motion of the neck.

SECONDARY OUTCOMES:
Infant/Toddler Sensory Profile | 1-12 months
  Infant/Toddler Sensory Profile; It will be used to evaluate sensory development. It is a questionnaire completed by the child's primary caregiver to collect information about sensory processing abilities. It is a questionnaire that questions the behavior and performance of a child between the ages of 0-3 (0-7 months and 7-36 months) regarding sensory processing. The test evaluates sensory processing in 6 different areas. These items; It consists of general, visual, auditory, vestibular, tactile and oral sensory processing. The caregiver evaluates the child's behavior on a 5-point scale. A score of one means "almost always" and a score of five means "almost never". The test score is evaluated in four test-specific groups: sensory sensitivity, sensory seeking, sensory avoidance, and low register.

CONTACTS AND LOCATIONS:
Overall Officials: Sinem ERTURAN, Principal Investigator — Study Principal Investigator
Locations (1):
- Rabia ZORLULAR, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Stellwagen L, Hubbard E, Chambers C, Jones KL. Torticollis, facial asymmetry and plagiocephaly in normal newborns. Arch Dis Child. 2008 Oct;93(10):827-31. doi: 10.1136/adc.2007.124123. Epub 2008 Apr 1. PMID 18381343
- [Result] Aarnivala HE, Valkama AM, Pirttiniemi PM. Cranial shape, size and cervical motion in normal newborns. Early Hum Dev. 2014 Aug;90(8):425-30. doi: 10.1016/j.earlhumdev.2014.05.007. Epub 2014 Jun 13. PMID 24951081
- [Result] Sargent B, Kaplan SL, Coulter C, Baker C. Congenital Muscular Torticollis: Bridging the Gap Between Research and Clinical Practice. Pediatrics. 2019 Aug;144(2):e20190582. doi: 10.1542/peds.2019-0582. PMID 31350358
- [Result] Hardgrib N, Rahbek O, Moller-Madsen B, Maimburg RD. Do obstetric risk factors truly influence the etiopathogenesis of congenital muscular torticollis? J Orthop Traumatol. 2017 Dec;18(4):359-364. doi: 10.1007/s10195-017-0461-z. Epub 2017 Jun 29. PMID 28664414